CLINICAL TRIAL: NCT01475253
Title: A Phase 2a Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study Evaluating Safety, Tolerability and Efficacy of LiRIS® in Women With Interstitial Cystitis Followed by an Open Label Extension
Brief Title: Double-Blind Placebo Controlled Study of Safety,Tolerability, and Efficacy of LiRIS® in Women With Interstitial Cystitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was not enrolled completely and was terminated.
Sponsor: Allergan (Industry)
Collaborators: TARIS Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAR-100-201
Record Dates: First submitted 2011-11-03; First posted 2011-11-21 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-08

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lidocaine Releasing Intravesical System (Experimental): Lidocaine Releasing Intravesical System (LiRIS®) is inserted into the bladder via cystoscopy on Study Day 0 and removed on Study Day 14. LiRIS releases lidocaine gradually during the 14 day indwelling period.
  Interventions: Drug: Lidocaine Releasing Intravesical System - LiRIS®
- LiRIS containing inactive substance only (Placebo Comparator): LiRIS Placebo is inserted into the bladder via cystoscopy on study Day 0 and removed via cystoscopy on study Day 14.
  Interventions: Other: LiRIS Placebo
- Cystoscopy Procedure (Sham Comparator): No intervention. Cystoscopy procedure is performed on study Day 0 and study Day 14 to mimick active and placebo study arms without insertion of Investigational Product into the bladder.
  Interventions: Procedure: Sham Cystoscopy Procedure

INTERVENTIONS:
Drug: Lidocaine Releasing Intravesical System - LiRIS® — Lidocaine Releasing Intravesical System (LiRIS®) is inserted into the bladder via cystoscopy on Study Day 0 and removed on Study Day 14. LiRIS releases lidocaine gradually during the 14 day indwelling period.
  Other Names: LiRIS® 400 mg; LiRIS® 400 mg (Active)
  Arms: Lidocaine Releasing Intravesical System
Other: LiRIS Placebo — LiRIS Placebo contains inactive substance only; LiRIS Placebo is inserted into the bladder via cystoscopy on study Day 0 and removed via cystoscopy on study Day 14.
  Other Names: LiRIS® 400 mg Placebo
  Arms: LiRIS containing inactive substance only
Procedure: Sham Cystoscopy Procedure — Cystoscopy procedure only; no investigational product is inserted/removed from the bladder.
  Other Names: Sham Comparator; Sham arm
  Arms: Cystoscopy Procedure

SUMMARY:
The purpose of this study is to determine if LiRIS®, an investigational drug-delivery system, is safe, tolerable and effective in women with Interstitial Cystitis. LiRIS® is inserted into the bladder via cystoscopy , remains in the bladder for 14 days, and is removed via cystoscopy.

DETAILED DESCRIPTION:
The study is conducted in 2 parts - a randomized, blinded part in which patients are randomly assigned to one of 3 possible arms (LiRIS® - contains lidocaine), LiRIS Placebo (LiRIS with inactive substance) or Sham(Insertion procedure only with neither LiRIS nor LiRIS Placebo), followed by an open extension part in which all patients are assigned to receive LiRIS® (with lidocaine). In part 1 of the study, treatment is managed in a double-blind manner for LiRIS® and LiRIS Placebo arms; and in a single-blind manner for the Sham arm (e.g.,the study doctor will know the treatment assignment for patients assigned to Sham).

All patients who complete part 1 of the study have the option to enter the extension.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 and over
* Diagnosed with Interstitial Cystitis as defined by protocol
* Able and willing to complete questionnaires and diary
* Able to comply with visit schedule including Day 14 Removal visit
* Completion of blinded study prior to enrolling in unblinded part of study

Exclusion Criteria:

* Pregnant or lactating women
* Bladder or urethra anatomical feature that would prevent the safe indwelling or insertion of the investigational product
* History or presence of any condition that would make it difficult to evaluate symptoms
* Did not complete blinded study (unblinded part of study only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Nickel, MD, Principal Investigator — Queen's University/Kingston General Hospital/Ontario Canada
Locations (29):
- United States (27):
  - Clinical Trials of Arizona, Glendale, Arizona
  - Citrus Valley Medical Research, Inc, Glendora, California
  - Stanford University Department of Urology, Stanford, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Grove Hill Clinical Research, New Britain, Connecticut
  - Manatee Medical Research Institute, LLC, Bradenton, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Center, Meridian, Idaho
  - First Urology, Jeffersonville, Indiana
  - Regional Urology LLC, Shreveport, Louisiana
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Bay State Clinical Trials, Inc, Watertown, Massachusetts
  - Female Pelvic Medicine & Urogynecology, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - CRC of Jackson and Southeast Urogynecology, Jackson, Mississippi
  - Sheldon Freedman, MD Ltd, Las Vegas, Nevada
  - Arthur Smith Institute for Urology, New Hyde Park, New York
  - University of Rochester, Department of Urology, Rochester, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Wake Forest University Health Sciences Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Penn. Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina Urology Ambulatory Care, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Integrity Medical Research, Mountlake Terrace, Washington
- Canada (2):
  - Pacific Urological Research, Victoria, British Columbia
  - Centre for Applied Urologic Research/Kingston General Hospital, Kingston, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited by clinical centers that saw subjects meeting eligibility criteria and were capable of undergoing cystoscopy per protocol specifications. The first subject was enrolled 28 November 2011.
Pre-assignment Details: In addition to meeting all protocol defined inclusion/exclusion criteria, participants were required to be females with a confirmed diagnosis of moderate to severe Interstitial Cystitis (IC) according to the 1987 National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) symptom severity criteria (modified to exclude cystometry).
Groups:
- LiRIS® 400 mg - Randomized Study: LiRIS® 400 mg, a non-resorbable intravesical drug-device combination investigational product that contains 400 mg of lidocaine, was inserted into the bladder using a standard cystoscopic procedure on Baseline Study Day 0 and was removed from the bladder on Day 14.
- LiRIS® Placebo-Randomized Study: LiRIS® Placebo, the matching placebo for the LiRIS® investigational product containing lactose as the drug surrogate, was inserted into the bladder using a standard cystoscopic procedure on Baseline Study Day 0 and was removed from the bladder on Day 14.
- Sham Cystoscopic Procedure-Randomized Study: Single-blinded "sham" arm of subjects who underwent cystoscopic insertion and retrieval procedures without any placement or removal of investigational product or placebo.
- LiRIS® 400 mg - Open Label Extension: LiRIS® 400 mg is a non-resorbable intravesical drug-device combination investigational product that contains 400 mg of lidocaine. All subjects who completed the randomized study had the option to enter the open label extension.
Period: Randomized, Blinded Study
Arm/Group | LiRIS® 400 mg - Randomized Study | LiRIS® Placebo-Randomized Study | Sham Cystoscopic Procedure-Randomized Study | LiRIS® 400 mg - Open Label Extension
Started | 47 | 46 | 11 | 0
Completed | 45 | 45 | 11 | 0
Not Completed | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Open Label Extension
Arm/Group | LiRIS® 400 mg - Randomized Study | LiRIS® Placebo-Randomized Study | Sham Cystoscopic Procedure-Randomized Study | LiRIS® 400 mg - Open Label Extension
Started | 0 | 0 | 0 | 56
Completed | 0 | 0 | 0 | 56
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LiRIS® 400 Mg-Randomized Study: LiRIS® 400 mg, a non-resorbable intravesical drug-device combination investigational product that contains 400 mg of lidocaine, was inserted into the bladder using a standard cystoscopic procedure on Baseline Study Day 0 and was removed from the bladder on Day 14.
- Total: Total of all reporting groups
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study | Sham Cystoscopic Procedure-Randomized Study | Total
Number analyzed (Participants) | 47 | 46 | 11 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 42 | 39 | 11 | 92
  >=65 years | 4 | 7 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (14.76) | 45.9 (15.85) | 38.1 (12.90) | 44.4 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 11 | 104
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 11 | 99
  Canada | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Responders Using the Global Response Assessment (GRA)
Description: Participants assessed their response to treatment using a seven item scale from Markedly improved to Markedly worse. A responder was defined as a participant who rated their symptoms as either Moderately or Markedly improved.
Time Frame: Baseline, Days 7, 14, 28 and 42
Population: Complete IDMC Population included all participants with available IDMC data. As per protocol, efficacy analyses were not performed for the Sham Cytoscopic Procedure-Randomized Study Arm/Group.
Measure: Number; unit: Percentage of Responders
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 42 | 40
Percentage of Responders
  Day 7 | 24 | 18
  Day 14 | 17 | 20
  Day 28 | 7 | 25
  Day 42 | 12 | 21

2. Primary Outcome: Change From Baseline in Participant Reported Bladder Pain as Assessed by a Visual Analog Scale (VAS) at Day 7
Description: Participant reported symptom of bladder pain in the prior 24 hours using a 10 centimeter (cm) horizontal line Pain Visual Analog Scale recorded in a diary. Participants were instructed to to put a mark on the line at the point that best described their bladder pain with 0 (far left on the line) reflecting no pain and 10 (far right on the line) reflecting worse possible pain. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 7
Population: Independent Data Monitoring Committee (IDMC) Population included data reviewed by the IDMC prior to study suspension. As per protocol, efficacy analyses were not performed for the Sham Cytoscopic Procedure-Randomized Study Arm/Group.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 42 | 40
centimeters | -1.25 (2.45) | -0.84 (1.92)

3. Primary Outcome: Change From Baseline in Participant Reported Bladder Pain as Assessed by a Visual Analog Scale (VAS) at Day 14
Description: Participant reported symptom of bladder pain in the prior 24 hours using a 10 centimeter horizontal line Pain Visual Analog Scale recorded in a diary. Participants were instructed to to put a mark on the line at the point that best described their bladder pain with 0 (far left on the line) reflecting no pain and 10 (far right on the line) reflecting worse possible pain. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 42 | 40
centimeters | -0.81 (2.50) | -0.45 (2.45)

4. Primary Outcome: Change From Baseline in Participant Reported Bladder Pain as Assessed by a Visual Analog Scale (VAS) ay Day 28
Description: as for outcome 3
Time Frame: Baseline, Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 42 | 40
centimeters | -0.92 (2.36) | -1.36 (2.28)

5. Primary Outcome: Change From Baseline in Participant Reported Bladder Pain as Assessed by a Visual Analog Scale (VAS) at Day 42
Description: as for outcome 3
Time Frame: Baseline, Day 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 42 | 40
centimeters | -0.89 (2.58) | -1.40 (2.51)

6. Secondary Outcome: Change From Baseline in Urinary Urgency as Assessed by VAS
Description: Urinary urgency was defined as an immediate unstoppable urge to urinate which may be due to a sudden involuntary contraction of the muscular wall of the bladder and may be accompanied by discomfort in the bladder. Participants reported symptom of urinary urgency in the last 24 hours using a Urgency Visual Analogue Scale (VAS). The Urgency VAS consists of a 10 centimeter (cm) horizontal line with the words "No Urgency" (best) at the left end (0 cm) and the words "Urgency as bad as you can imagine" (worst) at the right end (10 cm). Participants were instructed to complete the Pain VAS by marking the spot on the line that corresponded to their urinary urgency. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 7, 14, 28 and 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 43 | 40
centimeters
  Change from Baseline at Day 7 | 0.66 (2.66) | -1.45 (2.69)
  Change from Baseline at Day 14 | -0.76 (3.14) | -1.00 (2.74)
  Change from Baseline at Day 28 | -1.01 (2.93) | -1.77 (2.70)
  Change from Baseline at Day 42 | -0.30 (2.01) | -0.84 (2.74)

7. Secondary Outcome: Change From Baseline in Voiding Frequency
Description: Participants recorded Voiding Frequency in a 72 hour voiding log at Day 7, 14, 28 and 42. Lower numbers of voiding frequency is the best. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 7, 14, 28 and 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 43 | 40
Voids
  Change from Baseline at Day 7 | -7.3 (12.6) | -1.1 (20.3)
  Change from Baseline at Day 14 | -8.8 (13.2) | -5.8 (13.1)
  Change from Baseline at Day 28 | -9.3 (15.9) | -8.4 (12.8)
  Change from Baseline at Day 42 | -9.8 (15.3) | -7.2 (13.2)

8. Secondary Outcome: Change Form Baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) Score
Description: Participants answered four questions about bladder/voiding symptoms over the past month. 2 questions were on a scale of 0=Not at all to 5=Almost always, 1 question on a scale of 0=Not at all to 5=5 or more times per night and 1 questions from 0=Not at all to 4=Almost always for a total possible score of 0 (best) to19 (worst). A negative change from Baseline indicates improvement
Time Frame: Baseline, Days 7, 14, 28 and 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 43 | 40
score on a scale
  Change from Baseline at Day 7 | -2.39 (3.18) | -2.00 (3.56)
  Change from Baseline at Day 14 | -2.02 (3.90) | -1.97 (3.82)
  Change from Baseline at Day 28 | -2.93 (3.83) | -2.87 (3.68)
  Change from Baseline at Day 42 | -2.83 (4.11) | -2.32 (3.64)

9. Secondary Outcome: Change From Baseline in Interstitial Cystitis Problem Index (ICPI) Score
Description: Participants answered four questions about how bothersome their symptoms were over the past month using a 5 point scale: 1=No problem to 4=Big problem for a total possible score of 0 (best) to 16 worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 7, 14, 28 and 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 43 | 40
score on a scale
  Change from Baseline at Day 7 | -2.24 (2.74) | -1.54 (2.97)
  Change from Baseline at Day 14 | -2.33 (2.92) | -1.62 (3.21)
  Change from Baseline at Day 28 | -2.98 (3.14) | -2.23 (3.26)
  Change from Baseline at Day 42 | -2.48 (3.09) | -1.58 (3.01)

10. Secondary Outcome: Percentage of Participants With Change From Baseline in Cystoscopic Examination Findings
Description: Cystoscopic examinations were performed at Baseline and Day 14. The investigator assessed the urethra and bladder for the following: visibility of ureters, stricture, erythema, presence and number of Hunner's lesion(s) and the extent of erythema. For sites with the capability, videography or high resolution digital photographs of the bladder were taken. The findings at Day 14 were compared to the findings at Baseline and were reported as Improvement, Worsening or No Change.
Time Frame: Baseline, Day 14
Population: Intent-to-treat population included all enrolled participants for whom the study insertion procedure on Baseline Randomized was initiated. As per protocol, efficacy analyses were not performed for the Sham Cytoscopic Procedure-Randomized Study Arm/Group.
Measure: Number; unit: percentage of participants
Arm/Group | LiRIS® 400 Mg-Randomized Study | LiRIS® Placebo-Randomized Study
Number analyzed (Participants) | 46 | 46
percentage of participants
  Bladder Mucosal Erythema:Improvement | 35 | 15
  Bladder Mucosal Erythema:Worsening | 13 | 11
  Bladder Mucosal Erythema:No Change | 50 | 70
  Bladder Mucosal Erythema:Not Done | 2 | 4
  Hunner's Lesions:Improvement | 2 | 9
  Hunner's Lesions:Worsening | 2 | 2
  Hunner's Lesions:No Change | 96 | 89
  Stricture:Improvement | 0 | 0
  Stricture:Worsening | 0 | 0
  Stricture:No Change | 100 | 100

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) reporting was collected from the time of Day of insertion through the duration of study participation (Randomized and Open Label phases).[Up to 18 Weeks]
Description: The Intent-to-treat population, all enrolled participants for whom the study insertion procedure was initiated, was used for all safety analyses and was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Groups:
- LiRIS® Placebo - Randomized Study: LiRIS® Placebo, the matching placebo for the LiRIS investigational product containing lactose as the drug surrogate, was inserted into the bladder using a standard cystoscopic procedure on Baseline Study Day 0 and was removed from the bladder on Day 14.
- Sham Cystoscopic Procedure - Randomized Study: Single-blinded "sham" arm of subjects who underwent cystoscopic insertion and retrieval procedures without any placement or removal of investigational product or placebo.
- LiRIS 400 mg - Open Label Extension: LiRIS® 400 mg is a non-resorbable intravesical drug-device combination investigational product that contains 400 mg of lidocaine.
  All subjects who completed the randomized study had the option to enter the open lable extension.
Arm/Group | LiRIS® 400 mg - Randomized Study | LiRIS® Placebo - Randomized Study | Sham Cystoscopic Procedure - Randomized Study | LiRIS 400 mg - Open Label Extension
Serious Adverse Events (participants affected / at risk) | 1/46 | 2/46 | 0/11 | 0/56
Other Adverse Events (participants affected / at risk) | 23/46 | 23/46 | 7/11 | 29/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LiRIS® 400 mg - Randomized Study (N=46) | LiRIS® Placebo - Randomized Study (N=46) | Sham Cystoscopic Procedure - Randomized Study (N=11) | LiRIS 400 mg - Open Label Extension (N=56)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis Interstitial (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LiRIS® 400 mg - Randomized Study (N=46) | LiRIS® Placebo - Randomized Study (N=46) | Sham Cystoscopic Procedure - Randomized Study (N=11) | LiRIS 400 mg - Open Label Extension (N=56)
Dysuria (Renal and urinary disorders) | 11 (13) | 7 (8) | 0 (0) | 9 (12)
Bladder Pain (Renal and urinary disorders) | 8 (9) | 11 (12) | 1 (1) | 9 (10)
Bladder Discomfort (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 7 (7) | 2 (2) | 1 (1) | 6 (6)
Urethral Pain (Renal and urinary disorders) | 4 (5) | 3 (5) | 0 (0) | 4 (4)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4) | 2 (2) | 1 (1) | 7 (8)
Micturition Urgency (Renal and urinary disorders) | 3 (4) | 4 (4) | 0 (0) | 1 (1)
Bladder Irritation (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Headache (General disorders) | 3 (3) | 3 (5) | 0 (0) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 3 (4) | 0 (0) | 3 (3)
Abdominal Pain (Lower) (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Urine Odor Abnormal (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urine Abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Bacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papilloma Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Vulvovaginal Candidiasis
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema Peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Triglycerides Increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
As per protocol, efficacy analyses were not performed for the Sham Cytoscopic Procedure-Randomized Study Arm/Group. Only safety analyses were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other